| Participation and Environment Measure-Plus (PEM-Plus) Care Planning Intervention |
|---|
| NCT Number: 03820011 |

Date: June 17, 2017

Aim 1 Statistical Plan:

Demographic and usability data were exported via REDCap, and an administrative dashboard for analyses. Demographic characteristics and YC-PEM summary scores were reported for each user. To address the main study question, usability estimates were derived for the total study sample, according to technical effectiveness (PEM+ min-max and mean percent completion rate, mean completion time, and mean task difficulty rating), and USE summary scores (mean and range) for ease of use, ease of learning, and user satisfaction.

## Aim 2 Statistical Plan:

All analyses were completed on the total sample and age subgroups (0-3 years, 4-5 years) using SPSS 24.0. The primary study aim was to assess for PEM+ feasibility and acceptability. To assess for PEM+ feasibility, retention rate, median completion time of first iteration, median completion time of subsequent interactions, and use of tiered support were reported. To assess for PEM+ acceptability, total scores were reported as means with standard deviations. Additionally, open-ended responses were independently coded by four research team members to sort caregiver feedback regarding the acceptability of PEM+ into categories.

As a secondary aim, preliminary effects mean self-efficacy item scores were calculated and Pearson correlations were used to ascertain associations between proportion of care plans created, relative to areas of desired change, with caregiver self-efficacy scores.